CLINICAL TRIAL: NCT02677025
Title: Seek, Test, Treat, & Retain Pilot for Out of School Teens at Risk in Cape Town
Brief Title: Young Women's Health CoOp (Cooperative) in Cape Town
Acronym: YWHC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA032061 (NIH)
Record Dates: First submitted 2016-01-19; First posted 2016-02-09 (Estimated); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: HIV; Substance Abuse
Keywords: HIV; Sexual Risk; Sexually Transmitted Diseases; Substance Abuse; Violence and Victimization
MeSH Terms: conditions — Substance-Related Disorders; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Young Women's Health CoOp (YWHC) (Experimental): This is an adapted behavioral intervention for young women in Cape Town South Africa who dropped out of school, who use alcohol and other drugs and are at risk for HIV.
  Interventions: Behavioral: Young Women's Health CoOp (YWHC)
- HIV Counseling/Testing (Active Comparator): Provide age and gender appropriate standard HIV counseling and testing.
  Interventions: Behavioral: HIV Counseling/Testing

INTERVENTIONS:
Behavioral: Young Women's Health CoOp (YWHC) — Participants in this group will participate in two workshops of the young woman-focused intervention about HIV/STIs (sexually transmitted infections), sexual behaviors, alcohol and other drug use, violence, communication skills, and other issues. Participants will develop personalized risk reduction action plans at the end of each workshop session.
  Arms: Young Women's Health CoOp (YWHC)
Behavioral: HIV Counseling/Testing — Participants will be tested for HIV and if positive will receive counseling in accordance with national standards.
  Arms: HIV Counseling/Testing

SUMMARY:
This supplement study is an adaptation of the larger NIH-funded parent study, the Women's Health CoOp+, which tests a combination biobehavioral HIV prevention approach to enhance standard HIV testing practices for alcohol and drug (AOD)-using women across the city of Pretoria, South Africa. The current supplemental study seeks to reach AOD-using female adolescents who experience the greatest burden of new HIV infections and are currently underserved by HIV and drug-treatment programs in Cape Town, South Africa and test the validation of both the instrument and adapted intervention.

DETAILED DESCRIPTION:
This study is testing and validating both the revised instrument and adapted intervention through a small pilot trial where a cluster randomized design is used to recruit 100 participants through snowball sampling by community to either the YWHC condition or standard HIV Counseling and Testing (HCT); collect biological specimens to screen for recent drug use, pregnancy and HIV infection and provide referrals for care to resources; conduct process evaluation measures for satisfaction and a 1-month follow-up post-intervention interview assessing the feasibility and preliminary efficacy of conducting this intervention among vulnerable young women and linking them to care.

Young women from disadvantaged communities in Cape Town who have dropped out of school and who use AODs are highly vulnerable to physical victimization (violence and sexual victimization) from any perpetrator, including main sexual partners and drug-related sexual risks for HIV. Yet these vulnerable young women remain underserved by current HIV and drug treatment programs in the region, even though they are experiencing the greatest burden of new HIV infections in the country. The adapted Young Women's Health CoOp (YWHC) intervention has a high likelihood of wider implementation, sustainability, and a significant public health impact by reducing the exceedingly high HIV incidence amongst the most vulnerable populations in South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Female, 16 to 21 years of age
* Dropped out of school for at least 6 months
* Currently dropped out of school
* Have not completed matric or N 3 certificate
* Have used at least one drug (which can include alcohol) at least weekly in the past 90 days
* Report unprotected sex with a male partner in the last 90 days
* Able to provide informed assent to participate or informed consent if at least 18 years old
* Live in a targeted community Delft, Khayelitsha, or Mfuleni

Exclusion Criteria:

• Have been a part of formative activities

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Unprotected intercourse among women | One month post-intervention
  Percentages of condom use at last sex

SECONDARY OUTCOMES:
Alcohol use | One month post-intervention
  Frequency of alcohol use in past 30 days measured by RRBA (Revised Risk Behavior Assessment) and breath test
Alcohol use | One month post-intervention
  Frequency of alcohol use in past 30 days measured by breath test
Substance use | One month post-intervention
  Use of benzodiazepines, cocaine, methamphetamine, MDMA (methylenedioxymethamphetamine), marijuana and/or mandrax as determined by PRBA (Pretoria Risk Behavior Assessment)
Substance use | One month post-intervention
  Use of benzodiazepines, cocaine, methamphetamine, MDMA (methylenedioxymethamphetamine), marijuana and/or mandrax as determined by self-report
Victimization | One month post-intervention
  Percentages of young women who report being beaten in the previous 30 days
Victimization | One month post-intervention
  Percentages of young women who report being attacked with a weapon in the previous 30 days
Victimization | One month post-intervention
  Percentages of young women who report being forced to have sex in the previous 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Felicia Browne, ScD, Principal Investigator — RTI International
Locations (1):
- RTI International, Research Triangle Park, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
After the main findings are published, we welcome other researchers who want to analyze the data in other ways. Before this time, however, we anticipate establishing a publication plan that involves other researchers and institutions. Analytic data sets will be prepared in accordance with the "Privacy Rule" of the Health Insurance Portability and Accountability Act (HIPAA; http://www.hhs.gov/ocr/) as "limited data sets" in which names and other personal health identifiers are removed, birthdays have been converted to age at intake, and other dates have been changed to be days before or after the date of intake.

REFERENCES:
- [Derived] Carney T, Browne FA, Myers B, Kline TL, Howard B, Wechsberg WM. Adolescent female school dropouts who use drugs and engage in risky sex: effects of a brief pilot intervention in Cape Town, South Africa. AIDS Care. 2019 Jan;31(1):77-84. doi: 10.1080/09540121.2018.1500008. Epub 2018 Jul 18. PMID 30021470